CLINICAL TRIAL: NCT06922032
Title: A Novel Auditory Application for Distraction in Pediatric Patients: A Pilot Feasibility and Acceptability Study
Brief Title: A Novel Auditory Application for Distraction in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 80354
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-07

CONDITIONS: Emotional Distress
Keywords: Game engagement; Awe; Procedural Distraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mystics Pets group (Experimental)
  Interventions: Device: Mystics Pet

INTERVENTIONS:
Device: Mystics Pet — Participants will receive the game intervention and be instructed to wear a Oculus Quest 2 headset (Meta, Inc., Menlo Park, CA) and participate in Mystic Pets software game (Stanford Chariot Program, Palo Alto, CA) that is specifically designed to promote overall distraction and emotional distress reduction.

SUMMARY:
This mixed-methods study seeks to evaluate the feasibility of Mystic Pets software and hardware within the pediatric population. This study will take place at Lucile Packard Children's Hospital (Stanford University, Palo Alto, CA).

DETAILED DESCRIPTION:
Hospitalized children often experience emotional distress related to medical procedures, unfamiliar environments, and limited control over their situations. Existing distraction techniques, such as traditional videos and gaming, often rely heavily on visual interfaces, which can be limiting in clinical contexts. Current immersive technology software and hardware for procedural distraction rely on partial to complete immersion in a computer-generated environment to the real world. While immersive technology can reduce emotional distress with distraction, some patients experience increased distress due to loss of visual connection with their surroundings and/or caregivers. Using a head-mounted device and hand-gesture inputs, Mystic Pets maintains visual contact with a person's surroundings while gameplay is advanced through audio input and hand-gestures.

This research will significantly contribute to the growing field of digital therapeutics by providing early-stage data on a novel, immersive technology tailored to pediatric clinical care. If proven feasible, Mystic Pets could expand the toolkit available for procedural distraction, enhance patient comfort, and reduce the reliance on pharmacological interventions for emotion distress management.

The study also aims to establish preliminary engagement and usability benchmarks to guide future development and deployment of similar technologies in hospital environments.

ELIGIBILITY:
Inclusion Criteria:

* Between 4-17 years
* English speaking participants

Exclusion Criteria:

* Legal guardian not present to obtain consent
* Child with hearing impairment
* Child with a significant neurological condition, or major developmental disability
* Child with facial abnormalities or injuries prohibiting use of headsets
* Nausea at the time of recruitment,
* A history of severe motion sickness,
* A history of seizures

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Mystics Pets, based on an unpublished focus group interview guide at the Department of Anesthesiology, Stanford University | immediately after intervention
  Participants will provide qualitative feedback on the acceptability and feasibility of the use of Mystics Pets. Example question will include: "Can you please tell me about your experience?"

SECONDARY OUTCOMES:
ISO Ergonomic scale | immediately after intervention
  The scale has 6 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
System Usability Scale (SUS) Score | immediately after intervention
  The scale has 10 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
Game Engagement score | immediately after intervention
  Game Engagement score measured by Game Engagement Questionnaire. The scale has 16 items. Scores ranges from 1-5 (1 = strongly disagree and 5 = strongly agree)
Evaluate awe levels measured by Awe Experience Scale - Short Form | immediately after intervention
  The scale has 12 items. Scores ranges from 1-7 (1 = strongly disagree and 7 = strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States